CLINICAL TRIAL: NCT05901909
Title: The Effect of the Education Program Based on the Precede-Proceed Model to the Caregivers of Stroke Home Care Patients on Care Giving Response, Perceived Social Support Level, and Patient Outcomes.
Brief Title: Training Given to Caregivers of Stroke Home Care Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Sumeyye Akcoban, Lecturer, Mustafa Kemal University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HMKU-KMY-SA-01
Record Dates: First submitted 2023-05-22; First posted 2023-06-13 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Stroke
Keywords: Stroke; Home Care Services; Caregivers; Social Support; Patient-Relevant Outcome
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: two groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stroke home care patient (No Intervention): Before applying the education program based on the Precede-Proceed Model to 70 individuals who care for stroke home care patients, the evaluation of the patients will be made with home visits. After the training is given to the caregivers, the first evaluation will be made at the 8th week in order to determine the change in patient results after the training is completed. In the 16th week after the completion of the training, a final evaluation will be made with home visits to determine the change in patient results.
- Individuals caring for stroke home care patients (Experimental): Before the training program based on the Precede-Proceed Model is applied to the 70 individuals who care for stroke home care patients, the evaluation of the caregivers will be made in the hospital meeting room. After the training is given to the caregivers, the first evaluation will be made at the 8th week in order to determine the changes in their caregiving reactions and social support perceptions after the training is completed. In the 16th week after the completion of the training, a final evaluation will be made in the hospital meeting room in order to determine the changes in caregiver reactions and social support perceptions.
  Interventions: Behavioral: Educational intervention based on the Precede-Proceed Model for individuals caring for stroke home care patients

INTERVENTIONS:
Behavioral: Educational intervention based on the Precede-Proceed Model for individuals caring for stroke home care patients — Home visits will be made to 70 stroke patients identified during the implementation phase of the research, and training based on the Precede-Proceed model will be given to 70 individuals who care for these patients in the meeting room of the hospital where the research will be conducted. In the research, pre-education evaluation will be collected at the hospital before the training for the caregivers and home visits for the patients. In the second stage, the training program planned for the caregivers will be implemented in the meeting room of the hospital. After the training program reaches all of the caregivers in the determined number, the first evaluation will be made for the caregivers and the patient in the 8th week after the training is over. The third stage is the 16th week after the completion of the training, and the final evaluation will be made for the patients and caregivers.
  Arms: Individuals caring for stroke home care patients

SUMMARY:
Although stroke home care patients receive various treatments, they generally continue their lives as semi-dependent or fully dependent. Considering that stroke patients are especially elderly individuals, it is seen that they receive home health services and need a caregiver. The caregiver feels themselves under a heavy burden due to the lack of knowledge and insufficient experience. In addition, the lack of social support levels and the lack of training in patient care cause negative effects on patient outcomes.

DETAILED DESCRIPTION:
The research will be carried out face-to-face with 70 stroke patients who receive health care from the home health services unit of a State Hospital and 70 individuals who care for these patients between July 2023 and December 2023. This study is a single-sample study with its own control group. During the implementation phase of the research, home visits will be made to the patients and training based on the Precede-Proceed model will be given to the individuals who care for the patients in the meeting room of the hospital where the research will be conducted. The collection of research data will take place in three stages. In the research, pre-education evaluation will be collected at the hospital before the training for the caregivers and home visits for the patients. In the second stage, the training program planned for the caregivers will be implemented in the meeting room of the hospital. After the training program reaches all of the caregivers in the determined number, the first evaluation will be made for the caregivers and the patient in the 8th week after the training is over. The third stage is the 16th week after the completion of the training, and the final evaluation will be made for the patients and caregivers. In the study, data will be collected using the individual caregiver personal information form, the caregiver response rating scale and the multidimensional perceived social support scale, and the patient personal information form for the patients. Statistical significance level will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who care for semi-dependent or fully dependent stroke home care patients who agree to participate in the study,
* No communication problems,
* Do not have any psychiatric disorders that will reduce the ability to comprehend and understand,
* Caregivers over the age of 18.
* Semi-dependent or fully dependent stroke home care patients,
* Adult patients,
* Patients whose legal guardians or who have agreed to participate in the research themselves,

Exclusion Criteria:

* The refusal of caregivers or patients to participate in the study,
* The caregiver ceases to provide care or the patient dies during the research,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Patient Evaluation Form | In the first week after the start of the study, home visits will be made and the patients will be evaluated through the patient evaluation form.
  It is intended to evaluate the following findings. In this evaluation form: Presence of urinary catheter ()yes ()no, the last date of admission to the health institution, the status of applying to the health institution due to infection recently ()yes ()no, presence of pressure sores in the patient ()no, ()stage 1, ()stage 2, ()stage 3, ()stage 4, the patient's diet ()oral ()enteral ()parenteral, presence of constipation-diarrhea in the patient ()yes ()no, presence of incontinence in the patient ()yes () no, dementia status ()yes ()no, risk of falling ()yes ()no
Patient Evaluation Form | After the training program reaches all of the caregivers in the determined number and the training is completed, the first evaluation will be made for the patient in the 8th week.
  It is intended to evaluate the following findings. In this evaluation form: Presence of urinary catheter ()yes ()no, the last date of admission to the health institution, the status of applying to the health institution due to infection recently ()yes ()no, presence of pressure sores in the patient ()no, ()stage 1, ()stage 2, ()stage 3, ()stage 4, the patient's diet ()oral ()enteral ()parenteral, presence of constipation-diarrhea in the patient ()yes ()no, presence of incontinence in the patient ()yes () no, dementia status ()yes ()no, risk of falling ()yes ()no
Patient Evaluation Form | It is the 16th week after the completion of the training, and the final evaluation will be made for the patients.
  It is intended to evaluate the following findings. In this evaluation form: Presence of urinary catheter ()yes ()no, the last date of admission to the health institution, the status of applying to the health institution due to infection recently ()yes ()no, presence of pressure sores in the patient ()no, ()stage 1, ()stage 2, ()stage 3, ()stage 4, the patient's diet ()oral ()enteral ()parenteral, presence of constipation-diarrhea in the patient ()yes ()no, presence of incontinence in the patient ()yes () no, dementia status ()yes ()no, risk of falling ()yes ()no

SECONDARY OUTCOMES:
Caregiver Response Rating Scale | The caregivers will be evaluated by using the Caregiver Response Evaluation Scale within the first week before the individuals who care for stroke home care patients are given training.
  The Caregiver Response Evaluation Scale is used in the primary care of patients with physical and mental disorders to provide self-evaluation of caregivers. The scale consists of 24 items and 5 sub-dimensions. The scale has a 5-point Likert type scoring. Positive items in the scale; 7, 13, 3, 15, 19 while negative items are 1, 2, 4, 5, 6, 8, 9, 10, 11, 12, 14, 16, 17, 18, 20, 21, 22, 23, 24' type. While scoring the positive items, the value of 1 is converted to 5, and the value of 5 is converted to 1 in the scoring. In the scoring (total score 24-120), the scores of the answers given to the statements in each sub-dimension are summed, Interruption of daily life (5-25), financial distress (3-15), lack of family support (5-25), and health problems (4- High scores in the 20) sub-dimensions indicate that the caregivers are more distressed, and a high score in the Self-worth (7-35) sub-dimension indicates that the caregivers are in good condition.
Caregiver Response Rating Scale | After the training based on the Precede-Proceed Model is given to the caregivers of stroke home care patients, the caregivers will be evaluated using the Caregiver Response Evaluation Scale at the end of the 8th week.
  The Caregiver Response Evaluation Scale is used in the primary care of patients with physical and mental disorders to provide self-evaluation of caregivers. The scale consists of 24 items and 5 sub-dimensions. The scale has a 5-point Likert type scoring. Positive items in the scale; 7, 13, 3, 15, 19 while negative items are 1, 2, 4, 5, 6, 8, 9, 10, 11, 12, 14, 16, 17, 18, 20, 21, 22, 23, 24' type. While scoring the positive items, the value of 1 is converted to 5, and the value of 5 is converted to 1 in the scoring. In the scoring (total score 24-120), the scores of the answers given to the statements in each sub-dimension are summed, Interruption of daily life (5-25), financial distress (3-15), lack of family support (5-25), and health problems (4- High scores in the 20) sub-dimensions indicate that the caregivers are more distressed, and a high score in the Self-worth (7-35) sub-dimension indicates that the caregivers are in good condition.
Caregiver Response Rating Scale | After the training based on the Precede-Proceed Model is given to the caregivers of stroke home care patients, the caregivers will be evaluated using the Caregiver Response Evaluation Scale at the end of the 16th week.
  The Caregiver Response Evaluation Scale is used in the primary care of patients with physical and mental disorders to provide self-evaluation of caregivers. The scale consists of 24 items and 5 sub-dimensions. The scale has a 5-point Likert type scoring. Positive items in the scale; 7, 13, 3, 15, 19 while negative items are 1, 2, 4, 5, 6, 8, 9, 10, 11, 12, 14, 16, 17, 18, 20, 21, 22, 23, 24' type. While scoring the positive items, the value of 1 is converted to 5, and the value of 5 is converted to 1 in the scoring. In the scoring (total score 24-120), the scores of the answers given to the statements in each sub-dimension are summed, Interruption of daily life (5-25), financial distress (3-15), lack of family support (5-25), and health problems (4- High scores in the 20) sub-dimensions indicate that the caregivers are more distressed, and a high score in the Self-worth (7-35) sub-dimension indicates that the caregivers are in good condition.
Multidimensional Scale of Perceived Social Support | Individuals who care for stroke home care patients will be evaluated by using the Multidimensional Scale of Perceived Social Support in the first week without training.
  It is a scale to determine the social support elements perceived by individuals. The scale, which consists of 12 items in total, is a 7-point Likert-type scale (1-7) arranged as "definitely no 1 2 3 4 5 6 7 absolutely yes". It has three subscales. Items 3.4.8.11 in the scale measure support from family, items 6.7.9.12 measure support from friends and items 1.2.5.10 measure support from a special person. The lowest score that can be obtained from the subscales is 4 and the highest score is 28. The lowest score to be obtained from all of them is 12 and the highest score is 84. A high score indicates high perceived social support.
Multidimensional Scale of Perceived Social Support | After the training based on the Precede-Proceed Model is given to the caregivers of stroke home care patients, the caregivers will be evaluated using the Multidimensional Scale of Perceived Social Support at the end of the 8th week.
  It is a scale to determine the social support elements perceived by individuals. The scale, which consists of 12 items in total, is a 7-point Likert-type scale (1-7) arranged as "definitely no 1 2 3 4 5 6 7 absolutely yes". It has three subscales. Items 3.4.8.11 in the scale measure support from family, items 6.7.9.12 measure support from friends and items 1.2.5.10 measure support from a special person. The lowest score that can be obtained from the subscales is 4 and the highest score is 28. The lowest score to be obtained from all of them is 12 and the highest score is 84. A high score indicates high perceived social support.
Multidimensional Scale of Perceived Social Support | After the training based on the Precede-Proceed Model is given to the caregivers of stroke home care patients, the caregivers will be evaluated using the Multidimensional Scale of Perceived Social Support at the end of the 16th week.
  It is a scale to determine the social support elements perceived by individuals. The scale, which consists of 12 items in total, is a 7-point Likert-type scale (1-7) arranged as "definitely no 1 2 3 4 5 6 7 absolutely yes". It has three subscales. Items 3.4.8.11 in the scale measure support from family, items 6.7.9.12 measure support from friends and items 1.2.5.10 measure support from a special person. The lowest score that can be obtained from the subscales is 4 and the highest score is 28. The lowest score to be obtained from all of them is 12 and the highest score is 84. A high score indicates high perceived social support.

CONTACTS AND LOCATIONS:
Overall Officials: SÜMEYYE AKÇOBAN, Principal Investigator — Mustafa Kemal University
Locations (1):
- Hatay Mustafa Kemal University, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akcoban S, Eskimez Z. Homecare patients' quality of life and the burden of family caregivers: a descriptive cross-sectional study. Home Health Care Serv Q. 2023 Jul-Sep;42(3):216-229. doi: 10.1080/01621424.2023.2177224. Epub 2023 Feb 12. PMID 36774648
- [Background] Langhorne P, Ramachandra S; Stroke Unit Trialists' Collaboration. Organised inpatient (stroke unit) care for stroke: network meta-analysis. Cochrane Database Syst Rev. 2020 Apr 23;4(4):CD000197. doi: 10.1002/14651858.CD000197.pub4. PMID 32324916
- [Background] Sezgin D, Esin MN. Effects of a PRECEDE-PROCEED model based ergonomic risk management programme to reduce musculoskeletal symptoms of ICU nurses. Intensive Crit Care Nurs. 2018 Aug;47:89-97. doi: 10.1016/j.iccn.2018.02.007. Epub 2018 Mar 31. PMID 29609839